CLINICAL TRIAL: NCT02576197
Title: A Double Blind, Randomized, Placebo-Controlled Intervention Study to Evaluate the Effectiveness and Safety of a Treatment With a Probiotic in Adult Patients Diagnosed With Mild to Moderate Plaque Psoriasis
Brief Title: Intervention Study to Evaluate a Probiotic in Mild to Moderate Psoriasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biopolis S.L. (Industry)
Collaborators: Korott, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PSO/PRO 2
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Psoriasis
Keywords: mild to moderate; probiotic
MeSH Terms: conditions — Psoriasis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): one capsule per day, containing the probiotic along with the patient's customary psoriasis treatment (excluding systemic treatments)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): one capsule per day, containing the placebo, along with the patient's customary psoriasis treatment (excluding systemic treatments)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — one capsule per day, containing the probiotic along with the patient's customary psoriasis treatment (excluding systemic treatments)
  Arms: Probiotic
Dietary Supplement: Placebo — one capsule per day, containing the placebo, along with the patient's customary psoriasis treatment (excluding systemic treatments)
  Arms: Placebo

SUMMARY:
This study evaluates the efficiency of a probiotic as a coadjuvant in the conventional treatment of mild to moderate plaque psoriasis. Half of the patients will receive the probiotic per os, while the other half will receive a placebo; all patients will continue with their regular psoriasis treatment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficiency of a probiotic in capsules as a coadjuvant in the conventional treatment of mild to moderate plaque psoriasis. The efficiency is measured as the reduction in the PASI score in the patients (18 to 70 years old) included in the study, with a mild to moderate plaque psoriasis treated exclusively with topic treatment in the moment of being included in the study. Apart from the PASI score reduction from the first visit to the end of the study, the ability to reduce the improvement time in those patients will be evaluated as well. Additionally, the following markers of systemic inflammation are also compared between both active and placebo branches: Tumor necrosis factor, Interferon-gamma, interleukines 1b, 12, 16 and 23.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis diagnosed at least a year before the beginning of the treatment.
* Mild to moderate Psoriasis with a PASI score higher than 6 with no new flare-up in the previous four week to the beginning of the treatment.
* Patients capable of giving their informed consent to their participation in the study
* For women in fertile age, a negative pregnancy test before the beginning of the treatment, and the use of active contraceptive methods is required

Exclusion Criteria:

* Patients suffering from Crohn disease, hepatic cirrhosis, morbid obesity, VIH-positive or any other active infection.
* The use of any systemic, oral or parenteral psoriasis treatment in the last three months.
* The use of any antibiotic, probiotic or/and prebiotic in the last two weeks.
* The use of natural product with proved efficiency on health (apart from multivitamin and multimineral products)
* Any hepatic, renal, endocrine, respiratory, neurologic or cardiovascular disease.
* Pregnancy and breastfeeding.
* Patients not being capable of giving their informed consent or not being capable of following the study conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with a PASI score reduction higher than 75% | twelve weeks
  Number of patients with a PASI score reduction higher than 75% from the basal value
Time to reach a reduction in the PASI score higher than 75% | twelve weeks
  time to reach a reduction in the PASI score higher than 75% in from the basal value

SECONDARY OUTCOMES:
Average time to reach the clinical remission | twelve weeks
  Average time to reach the clinical remission, with no activity (PASI score lower than 6) from the treatment beginning
Differences among any of the inflammation markers | twelve weeks
number of patients that remains in analytical remission | twelve weeks
  number of patients that remains in analytical remission (that is, that maintain said inflammation markers in normal values)
Number of patients with mild, moderate or severe adverse events | twelve weeks
  Number of patients with mild, moderate or severe adverse events attributable to regular treatment to psoriasis or to probiotic.
Number of patients with an improvement in the PGA score | Twelve weeks
  Number of patients with an improvement in the PGA score at the end of the study with regard of basal values

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Navarro-López, MD, Principal Investigator — Universidad Católica San Antonio de Murcia; Ana A Ramirez-Boscá, MD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Centro Dermatológico Estético de Alicante, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramirez-Bosca A, Navarro-Lopez V, Martinez-Andres A, Such J, Frances R, Horga de la Parte J, Asin-Llorca M. Identification of Bacterial DNA in the Peripheral Blood of Patients With Active Psoriasis. JAMA Dermatol. 2015 Jun;151(6):670-1. doi: 10.1001/jamadermatol.2014.5585. No abstract available. PMID 25760018
- [Background] Betsi GI, Papadavid E, Falagas ME. Probiotics for the treatment or prevention of atopic dermatitis: a review of the evidence from randomized controlled trials. Am J Clin Dermatol. 2008;9(2):93-103. doi: 10.2165/00128071-200809020-00002. PMID 18284263